CLINICAL TRIAL: NCT04504695
Title: Prediction of Patient-specific Outcomes After Interventional Neuroradiology Procedures
Acronym: PREDICTNRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: INTRADYS (Unknown)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0032
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Aneurysmal Disease; Stroke
Keywords: thrombectomy; aneurysm
MeSH Terms: conditions — Stroke; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombectomy group: Major patients requiring management for endovascular thrombosis
- Aneurysm group: Major patients requiring management for an intracranial aneurysm

SUMMARY:
Stroke is either an obstruction (ischemic stroke) or the rupture of a blood vessel in the brain (ruptured aneurysm). It can happen at any age in adults. Because of the risk of irreversible brain damage, it is an absolute medical emergency.

An ischemic stroke (stroke) is the result of a lack of oxygen supply to a part of the brain. It can be one of many causes of stroke as a result of a thrombosis (occlusion) of the internal carotid artery or a cerebral embolism (migration of a clot or debris of fatty deposits) from a carotid stenosis. In both cases part of the brain is less irrigated. There will then be a neurological deficit (paralysis) more or less important corresponding to the affected cerebral territory. The deficit may concern the whole hemicorps (hemiplegia) or a part of the body (upper or lower limb) and sometimes is associated with facial paralysis and/or language disorders.

A brain aneurysm occurs when the wall of an intracranial artery expands abnormally, creating a pocket of blood. It is often caused by weakness in the vascular tissue, but it can also occur later in life due to illness, head injury, oral contraceptives or certain lifestyle habits (smoking, excessive alcohol consumption). Sudden increases in pressure due to stress or strenuous exercise can serve as a trigger.

Interventional Neuroradiology (INR) is a medical specialty that manages stroke patients using imaging to perform the medical procedure and thereby limit openings and their associated risks. This specialty has a growing place in modern medicine.

In order to improve the quality of care, patient safety and functional outcomes, it is necessary to keep patient information. A database storing patient data from the NRI department will make it possible to track patients since their arrival at the Brest University Hospital. Thanks to this structured database, clinical studies will be facilitated, making it possible to advance knowledge of the pathology and its treatments.

From the bibliographical research, we can conclude as to the current state of the facts: there is currently no method for predicting the functional results of the interventional neuroradiologist's patient based on automated learning.

A strategy based on an innovation programme is therefore being implemented over several years, the first stage of which is the retrospective data study which was approved by the ethics committee on 12/09/2019 and the second stage is the prospective data study.

This innovation program requires the most complete and homogeneous data possible.

ELIGIBILITY:
Inclusion Criteria:

- Major patient carrying either a small or large, ruptured or unruptured aneurysm or a thrombectomy, with in both cases, a treatment procedure carried out in the interventional neuroradiology department of the Brest CHRU.

Exclusion Criteria:

* Age < 18 years old
* Incapacitated patients of full age (under guardianship or curatorship)
* Refusal to participate
* Follow-up impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient carrying either a small or large, ruptured or unruptured aneurysm or a thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-01-04 (Estimated); Study Completion 2025-01-04 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive factors | 24 months
  Number of predictive factors (pre- and intra-operative data) for the angiographic success of the procedure (intracranial aneurysm or thrombectomy).

SECONDARY OUTCOMES:
Clinical evolution | 24 months
  Clinical evolution was followed by the relevant clinical signs
Neurological evolution | 24 months
  Neurological evolution was followed by the neurologicsigns

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending five years following the princeps publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.